CLINICAL TRIAL: NCT03616405
Title: Efficacy and Safety of a 14-day Modified Sequential Therapy for Refractory Helicobacter Pylori Infection: a Pilot Study
Brief Title: Pilot Study of a 14-day Modified Sequential Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018SDU-QILU-G001
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Sequential Therapy; Rescue Treatment
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Tetracycline; Furazolidone; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14-day modified sequential therapy (Experimental): All the participants will go through a gastroscopy. Biopsy specimens will be taken for histologic assessment and rapid urease test. Two additional biopsy samples will be obtained from the antrum and body for bacterial culture and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment.
  Then, patients will receive a 14-day modified sequential therapy for the Helicobacter pylori eradication irrespective of antimicrobial susceptibility test results. The regimen contains rabeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by rabeprazole，amoxicillin, tetracycline and colloidal bismuth pectin for the second 7 days.
  Drugs: 1. rabeprazole 10mg bid for 14 days, 2. amoxicillin 1000mg bid for 14 days, 3. tetracycline 500mg qid for 14 days, 4. furazolidone 100mg tid for the firs 7 days, 5. colloidal bismuth pectin 200mg bid for the second 7 days.
  Interventions: Drug: rabeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days)

INTERVENTIONS:
Drug: rabeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days) — Patients will go through a gastroscopy and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day modified sequential therapy for the Helicobacter pylori eradication. The regimen contains rabeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by rabeprazole，amoxicillin, tetracycline and colloidal bismuth pectin for the second 7 days.

SUMMARY:
The purpose of this study is to assess efficacy of a 14-day sequential therapy for the rescue treatment of refractory Helicobacter pylori infection, and whether it is safe while maintaining an ideal eradication rates.

DETAILED DESCRIPTION:
Half of the world's population is infected with Helicobacter pylori. Strong evidence supports that H.pylori eradication is an effective approach to reduce the risk of developing gastric cancer. However, eradication rates of first-line therapy decreased over years due to the rapidly emerging antibiotic resistance of H. pylori worldwide. An ideal rescue therapeutic regimen to cure refractory H.pylori infection is currently warranted.

Traditional sequential therapy failed to achieve an ideal eradication rates (over>95%) as a third line treatment in the region with high antibiotic resistance. The investigator's study aims to evaluate the efficacy 14-day modified sequential therapy in the patients with two or more treatment failure, and whether the adverse effects of this new modified sequential therapy are tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with persistent H. pylori infection.
* Patients failed at least three different standard eradication therapies before. Previous standard eradication therapy was defined as a 10-day or 14-day quadruple regimen designed according to Maastricht V report.

Exclusion Criteria:

* Patients unable or unwilling to receive gastroscopy.
* Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastorectomy, acute GI bleeding and advanced gastric cancer.
* History of allergy to any of the drugs used in the study.
* Severe concomitant cardiovascular, respiratory, or endocrine diseases, clinically significant renal or hepatic disease, hematologic disorders and any other clinically significant medical condition that could increase risk.
* Currently pregnant or lactating.
* Severe neurologic or psychiatric disorders.
* Alcohol abuse or drug addiction.
* Patients with compliance lower than 90% in any previous treatment are not included.
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rates | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infection. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of adverse events happening | 6 months
  Common adverse events will be measured using a 8-point Likert scale, and patients rate their symptoms from 0 (none) to 8 (severe) during the treatment process.
The rate of improving dyspepsia symptoms after Helicobacter pylori eradication. | 6 months
  Dyspepsia symptoms will also be measured using a 8-point Likert scale
The rate of good compliance | 6 months
  Patients taken over 90% of drugs are considered to have a good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China